CLINICAL TRIAL: NCT06096389
Title: Effect of Acheta Domesticus Supplementation on Post-Exercise Muscle Recovery in Recreationally Active Male
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UM.TNC2/UMREC_2337
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Muscle Soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Maltodextrin (CHO) (Placebo Comparator): This group will be given isocaloric carbohydrate (maltodextrin)
  Interventions: Other: 100 Drop Jumps; Dietary Supplement: Carbohydrate supplementation
- Whey Protein Isolate (WIP) (Active Comparator): This group will receive whey protein isolate
  Interventions: Other: 100 Drop Jumps; Dietary Supplement: Whey supplementation
- House Cricket (HCP) (Experimental): This group will receive house cricket powder
  Interventions: Other: 100 Drop Jumps; Dietary Supplement: House cricket supplementation

INTERVENTIONS:
Other: 100 Drop Jumps — 100 drop jumps from 60 cm height. Divided into 5 sets of 20 reps
Dietary Supplement: Whey supplementation — Consume whey protein isolate based on subjects' daily protein intake
  Arms: Whey Protein Isolate (WIP)
Dietary Supplement: Carbohydrate supplementation — Consume carbohydrate (isocaloric to whey)
  Arms: Maltodextrin (CHO)
Dietary Supplement: House cricket supplementation — Consume defatted house cricket powder based on subjects' daily protein intake
  Arms: House Cricket (HCP)

SUMMARY:
The goal of this clinical trial is to test the effect of house cricket (Acheta domesticus) supplementation for strength recovery in recreationally active males. The main question[s] it aims to answer are: whether house cricket powder could improve strength recovery and whether house cricket powder could be an alternative to commonly used protein supplement. Participants will do exercise (100 drop jumps) to induce fatigue and then they will consume either isocaloric carbohydrate, whey protein isolate or defatted house cricket powder for 4 days. Their strength will be measured every 24 hours for 4 days in order to observe the recovery.

Researcher will compare house cricket powder with isocaloric carbohydrate to see if the strength recovery is faster in house cricket powder group

Researcher will compare house cricket powder with whey protein isolate to see if the strength recovery is comparable.

DETAILED DESCRIPTION:
Participants: recreationally active males Study type: double-blind randomized controlled trial

Supplement dose is tailored to each participant daily protein consumption. It aims to reach 1.4 g/kg body weight protein, hence participant is required to provide dietary record 3 days before the experiment and during the experiment. Subject will attend one familiarization 1 week before the experiment. During day one of the experiment, subject warmed up before the session. Then their baseline strength and jumping measurement will be taken. Afterwards, they will do 20 reps of drop jumps for 5 sets (each set separated by 2 minutes rest). Immediately after the exercise, they will consume either whey, house cricket or maltodextrin. 10 minutes afterwards, they will undergo another strength and jumping measurement. 24, 48 and 72 hours after the exercise, subject will come for strength and jumping post-test after consuming the supplement. They are also required to fill in a visual analogue scale and 7-points Likert scale form regarding their pain and soreness perception.

ELIGIBILITY:
Inclusion Criteria:

* 5-10 hours of exercise per week

Exclusion Criteria:

* smoking
* drinking alcohol
* history of surgical/medical procedure that could affect the study
* food allergy
* in medication
* have participated in similar studies before

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Recreationally active males
Enrollment: 39 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Strength | 72 hours
  Isokinetic knee extension and flexion, maximum knee isometric contraction
Power | 72 hours
  Countermovement jump, squat jump
Pain Perception | 72 hours
  10 cm visual analogue scale (min 0 = no soreness, max 10 = worst imaginable muscle soreness) & 7 Points Likert Scale (min 0 = no soreness, max 6 = a severe pain that limits my ability to move)

CONTACTS AND LOCATIONS:
Overall Officials: Ashril Yusof, PhD, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Sports and Exercise Sciences, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abaidia AE, Delecroix B, Leduc C, Lamblin J, McCall A, Baquet G, Dupont G. Effects of a Strength Training Session After an Exercise Inducing Muscle Damage on Recovery Kinetics. J Strength Cond Res. 2017 Jan;31(1):115-125. doi: 10.1519/JSC.0000000000001479. PMID 27227793
- [Background] Agriculture Organization of the United Nations, World Health Organization, & University, U. N. (2007). Protein and amino acid requirements in human nutrition : report of a joint FAO/WHO/UNU expert consultation. World Health Organization. https://apps.who.int/iris/handle/10665/43411
- [Background] Awobusuyi TD, Pillay K, Siwela M. Consumer Acceptance of Biscuits Supplemented with a Sorghum-Insect Meal. Nutrients. 2020 Mar 25;12(4):895. doi: 10.3390/nu12040895. PMID 32218250
- [Background] Baiano A. (2020). Edible insects: an overview on nutritional characteristics, safety, farming, production technologies, regulatory framework, and socio-economic and ethical implications. Trends in Food Science & Technology. 100:35-50
- [Background] Brogan, E. N., Park, Y. L., Matak, K. E., & Jaczynski, J. (2021). Characterization of protein in cricket (Acheta domesticus), locust (Locusta migratoria), and silk worm pupae (Bombyx mori) insect powders. Lwt-Food Science and Technology, 152, Article 112314. https://doi.org/10.1016/j.lwt.2021.112314
- [Background] Brown MA, Stevenson EJ, Howatson G. Whey protein hydrolysate supplementation accelerates recovery from exercise-induced muscle damage in females. Appl Physiol Nutr Metab. 2018 Apr;43(4):324-330. doi: 10.1139/apnm-2017-0412. Epub 2017 Nov 6. PMID 29106812
- [Background] Borgenvik M, Apro W, Blomstrand E. Intake of branched-chain amino acids influences the levels of MAFbx mRNA and MuRF-1 total protein in resting and exercising human muscle. Am J Physiol Endocrinol Metab. 2012 Mar 1;302(5):E510-21. doi: 10.1152/ajpendo.00353.2011. Epub 2011 Nov 29. PMID 22127230
- [Background] Buckley JD, Thomson RL, Coates AM, Howe PR, DeNichilo MO, Rowney MK. Supplementation with a whey protein hydrolysate enhances recovery of muscle force-generating capacity following eccentric exercise. J Sci Med Sport. 2010 Jan;13(1):178-81. doi: 10.1016/j.jsams.2008.06.007. Epub 2008 Sep 2. PMID 18768358
- [Background] Buford TW, Kreider RB, Stout JR, Greenwood M, Campbell B, Spano M, Ziegenfuss T, Lopez H, Landis J, Antonio J. International Society of Sports Nutrition position stand: creatine supplementation and exercise. J Int Soc Sports Nutr. 2007 Aug 30;4:6. doi: 10.1186/1550-2783-4-6. No abstract available. PMID 17908288
- [Background] Abbott W, Brett A, Cockburn E, Clifford T. Presleep Casein Protein Ingestion: Acceleration of Functional Recovery in Professional Soccer Players. Int J Sports Physiol Perform. 2019 Mar 1;14(3):385-391. doi: 10.1123/ijspp.2018-0385. Epub 2019 Feb 17. PMID 30204517
- [Background] Cooke MB, Rybalka E, Stathis CG, Cribb PJ, Hayes A. Whey protein isolate attenuates strength decline after eccentrically-induced muscle damage in healthy individuals. J Int Soc Sports Nutr. 2010 Sep 22;7:30. doi: 10.1186/1550-2783-7-30. PMID 20860817
- [Background] Cormack SJ, Newton RU, McGuigan MR, Doyle TL. Reliability of measures obtained during single and repeated countermovement jumps. Int J Sports Physiol Perform. 2008 Jun;3(2):131-44. doi: 10.1123/ijspp.3.2.131. PMID 19208922
- [Background] de Matos FM, Novelli PK, de Castro RJS. Enzymatic hydrolysis of black cricket (Gryllus assimilis) proteins positively affects their antioxidant properties. J Food Sci. 2021 Feb;86(2):571-578. doi: 10.1111/1750-3841.15576. Epub 2021 Jan 12. PMID 33438276
- [Background] Eddens L, Browne S, Stevenson EJ, Sanderson B, van Someren K, Howatson G. The efficacy of protein supplementation during recovery from muscle-damaging concurrent exercise. Appl Physiol Nutr Metab. 2017 Jul;42(7):716-724. doi: 10.1139/apnm-2016-0626. Epub 2017 Feb 15. PMID 28199799
- [Background] Etheridge T, Philp A, Watt PW. A single protein meal increases recovery of muscle function following an acute eccentric exercise bout. Appl Physiol Nutr Metab. 2008 Jun;33(3):483-8. doi: 10.1139/H08-028. PMID 18461101
- [Background] Hansen M, Bangsbo J, Jensen J, Bibby BM, Madsen K. Effect of whey protein hydrolysate on performance and recovery of top-class orienteering runners. Int J Sport Nutr Exerc Metab. 2015 Apr;25(2):97-109. doi: 10.1123/ijsnem.2014-0083. Epub 2014 Jul 14. PMID 25029703
- [Background] Hermans WJH, Senden JM, Churchward-Venne TA, Paulussen KJM, Fuchs CJ, Smeets JSJ, van Loon JJA, Verdijk LB, van Loon LJC. Insects are a viable protein source for human consumption: from insect protein digestion to postprandial muscle protein synthesis in vivo in humans: a double-blind randomized trial. Am J Clin Nutr. 2021 Sep 1;114(3):934-944. doi: 10.1093/ajcn/nqab115. PMID 34020450
- [Background] Hilkens L, De Bock J, Kretzers J, Kardinaal AFM, Floris-Vollenbroek EG, Scholtens PAMJ, Horstman AMH, van Loon LJC, van Dijk JW. Whey protein supplementation does not accelerate recovery from a single bout of eccentric exercise. J Sports Sci. 2021 Feb;39(3):322-331. doi: 10.1080/02640414.2020.1820184. Epub 2020 Oct 5. PMID 33012216
- [Background] Kreider RB, Campbell B. Protein for exercise and recovery. Phys Sportsmed. 2009 Jun;37(2):13-21. doi: 10.3810/psm.2009.06.1705. PMID 20048505
- [Background] Kritikos S, Papanikolaou K, Draganidis D, Poulios A, Georgakouli K, Tsimeas P, Tzatzakis T, Batsilas D, Batrakoulis A, Deli CK, Chatzinikolaou A, Mohr M, Jamurtas AZ, Fatouros IG. Effect of whey vs. soy protein supplementation on recovery kinetics following speed endurance training in competitive male soccer players: a randomized controlled trial. J Int Soc Sports Nutr. 2021 Mar 16;18(1):23. doi: 10.1186/s12970-021-00420-w. PMID 33726784
- [Background] Navarro Del Hierro J, Gutierrez-Docio A, Otero P, Reglero G, Martin D. Characterization, antioxidant activity, and inhibitory effect on pancreatic lipase of extracts from the edible insects Acheta domesticus and Tenebrio molitor. Food Chem. 2020 Mar 30;309:125742. doi: 10.1016/j.foodchem.2019.125742. Epub 2019 Oct 25. PMID 31704068
- [Background] Nino MC, Reddivari L, Ferruzzi MG, Liceaga AM. Targeted Phenolic Characterization and Antioxidant Bioactivity of Extracts from Edible Acheta domesticus. Foods. 2021 Sep 28;10(10):2295. doi: 10.3390/foods10102295. PMID 34681345
- [Background] Oonincx DG, van Itterbeeck J, Heetkamp MJ, van den Brand H, van Loon JJ, van Huis A. An exploration on greenhouse gas and ammonia production by insect species suitable for animal or human consumption. PLoS One. 2010 Dec 29;5(12):e14445. doi: 10.1371/journal.pone.0014445. PMID 21206900
- [Background] Orkusz A. Edible Insects versus Meat-Nutritional Comparison: Knowledge of Their Composition Is the Key to Good Health. Nutrients. 2021 Apr 6;13(4):1207. doi: 10.3390/nu13041207. PMID 33917531
- [Background] Osimani, A., Milanović, V., Cardinali, F., Roncolini, A., Garofalo, C., Clementi, F., Pasquini, M., Mozzon, M., Foligni, R., Raffaelli, N., Zamporlini, F., & Aquilanti, L. (2018). Bread enriched with cricket powder (Acheta domesticus): A technological, microbiological and nutritional evaluation. Innovative Food Science & Emerging Technologies, 48, 150-163. https://doi.org/https://doi.org/10.1016/j.ifset.2018.06.007
- [Background] Paul, A., Frederich, M., Megido, R. C., Alabi, T., Malik, P., Uyttenbroeck, R., Francis, F., Blecker, C., Haubruge, E., Lognay, G., & Danthine, S. (2017). Insect fatty acids: A comparison of lipids from three Orthopterans and Tenebrio molitor L. larvae. Journal of Asia-Pacific Entomology, 20(2), 337-340. https://doi.org/https://doi.org/10.1016/j.aspen.2017.02.001
- [Background] Placentino U, Sogari G, Viscecchia R, De Devitiis B, Monacis L. The New Challenge of Sports Nutrition: Accepting Insect Food as Dietary Supplements in Professional Athletes. Foods. 2021 May 18;10(5):1117. doi: 10.3390/foods10051117. PMID 34070020
- [Background] Stull VJ, Finer E, Bergmans RS, Febvre HP, Longhurst C, Manter DK, Patz JA, Weir TL. Impact of Edible Cricket Consumption on Gut Microbiota in Healthy Adults, a Double-blind, Randomized Crossover Trial. Sci Rep. 2018 Jul 17;8(1):10762. doi: 10.1038/s41598-018-29032-2. PMID 30018370
- [Background] Tang JE, Moore DR, Kujbida GW, Tarnopolsky MA, Phillips SM. Ingestion of whey hydrolysate, casein, or soy protein isolate: effects on mixed muscle protein synthesis at rest and following resistance exercise in young men. J Appl Physiol (1985). 2009 Sep;107(3):987-92. doi: 10.1152/japplphysiol.00076.2009. Epub 2009 Jul 9. PMID 19589961
- [Background] Tipton KD, Elliott TA, Cree MG, Wolf SE, Sanford AP, Wolfe RR. Ingestion of casein and whey proteins result in muscle anabolism after resistance exercise. Med Sci Sports Exerc. 2004 Dec;36(12):2073-81. doi: 10.1249/01.mss.0000147582.99810.c5. PMID 15570142
- [Background] Trommelen J, van Loon LJ. Pre-Sleep Protein Ingestion to Improve the Skeletal Muscle Adaptive Response to Exercise Training. Nutrients. 2016 Nov 28;8(12):763. doi: 10.3390/nu8120763. PMID 27916799
- [Background] Udomsil, N., Imsoonthornruksa, S., Gosalawit, C., & Ketudat-Cairns, M. (2019). Nutritional values and functional properties of house cricket (Acheta domesticus) and field cricket (Gryllus bimaculatus). Food Science and Technology Research, 25(4), 597-605. https://doi.org/10.3136/fstr.25.597
- [Background] van Huis, A., van Itterbeeck, J., Klunder, H., Mertens, E., Halloran, A., Muir, G., Vantomme, P. (2013). Edible insects: future prospect for food and feed security. Food and Agriculture Organization of the United Nations.
- [Background] Vangsoe MT, Joergensen MS, Heckmann LL, Hansen M. Effects of Insect Protein Supplementation during Resistance Training on Changes in Muscle Mass and Strength in Young Men. Nutrients. 2018 Mar 10;10(3):335. doi: 10.3390/nu10030335. PMID 29534456
- [Background] Vangsoe MT, Thogersen R, Bertram HC, Heckmann LL, Hansen M. Ingestion of Insect Protein Isolate Enhances Blood Amino Acid Concentrations Similar to Soy Protein in A Human Trial. Nutrients. 2018 Sep 22;10(10):1357. doi: 10.3390/nu10101357. PMID 30248987
- [Background] Wilborn CD, Taylor LW, Outlaw J, Williams L, Campbell B, Foster CA, Smith-Ryan A, Urbina S, Hayward S. The Effects of Pre- and Post-Exercise Whey vs. Casein Protein Consumption on Body Composition and Performance Measures in Collegiate Female Athletes. J Sports Sci Med. 2013 Mar 1;12(1):74-9. eCollection 2013. PMID 24149728
- [Background] Witard OC, Jackman SR, Kies AK, Jeukendrup AE, Tipton KD. Effect of increased dietary protein on tolerance to intensified training. Med Sci Sports Exerc. 2011 Apr;43(4):598-607. doi: 10.1249/MSS.0b013e3181f684c9. PMID 20798660